CLINICAL TRIAL: NCT03733054
Title: Understanding Prosthetic Needs and Outcomes in Women Veterans With Amputation
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: A2797-R
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Amputation
Keywords: female; Veterans; Quality of life; Prostheses; Lower extremity amputation; Surveys and questionnaires; electronic health records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — No biospecimens are being collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Men: Men with lower limb amputation
- Women: Women with lower limb amputation

SUMMARY:
The proportion of US Veterans who are women is currently at its highest point in history and is projected to continue increasing. Nonetheless, the literature regarding prosthetic and functional outcomes in women Veterans with lower extremity amputation (LEA) is nearly non-existent. Research in other healthcare systems indicates the presence of concerning gender differences in both prosthetic outcomes and functional mobility, with women being less likely to be prescribed a prosthesis, less likely to use it, and more likely to be dissatisfied than men. This mixed-methods study will use VA administrative data, qualitative interviews, and a patient survey to characterize women Veterans' outcomes as well as compare them to those of male Veterans, resulting in the largest study to date on women Veterans with LEA. Data from this rigorous evaluation will inform clinical care by identifying intervention targets to improve prosthetic and functional outcomes for this understudied population.

DETAILED DESCRIPTION:
Background: The VA has a long history of developing and providing state-of-the-art prosthetic technology and rehabilitation services for Veterans with lower extremity amputations (LEA). Despite VA's goal to provide patient-centered, gender-sensitive care to all Veterans, prosthetics research in VA has mainly included and focused on the needs of men. Women are the fastest growing demographic in VA, and VA currently provides care to over 1,200 women with a major LEA. That number will likely increase as the number of women Veterans, currently at its highest point in history, is expected to continue rising. Primary goals of rehabilitation following a major LEA include successfully fitting a prosthesis and providing training to use the prosthesis to achieve functional mobility. Greater prosthesis use is associated with improved mobility, functioning, and independence as well as better quality of life. Thus, identifying the extent to which women achieve functional mobility through prostheses that fit them and meet their needs is critical to ensure that VA is providing excellent and equitable care. Accordingly, the goal of this research is to provide information that will improve clinical care for women Veterans with LEA.

Objectives: The objectives of this study are to: 1) characterize prosthetic prescription rates, prosthetic-device types, time to prescription, and their correlates among women with major LEA as well as evaluate gender differences in these outcomes using administrative data; 2) identify barriers and facilitators to achieving successful functional mobility, factors impacting prosthetic use and satisfaction, and needs and preferences related to prostheses among women with major LEA who were prescribed a prosthesis using qualitative interviews; and 3) characterize prosthetic use, prosthetic satisfaction, functional mobility, and health-related quality of life and their correlates among women as well as evaluate gender differences in these outcomes using survey data.

Methods: To achieve these objectives, the investigators will capitalize on VA's extensive electronic medical record data, including the Corporate Data Warehouse (Aim 1), qualitative interviews (Aim 2) and a quantitative survey (Aim 3) with Veterans with LEA. Both administrative data and the survey will include women and men, to characterize women overall and in comparison to men. The investigators will determine which patients have received prescriptions for definitive prostheses by linking procedure data related to amputations and prosthetics data (which are all available within the Corporate Data Warehouse); other outcomes will be assessed via survey. For Aim 2, the investigators will conduct semi-structured telephone interviews with a sample of women with a major LEA who were prescribed a prosthesis. Aim 3 will involve a self-administered mailed survey that will permit us to characterize prosthetic use, prosthetic satisfaction, functional mobility, and health-related quality of life and evaluate clinical, social/environmental, and prosthetist/prostheses-related factors as potential determinants of outcomes among women as well as potential mediators that explain observed gender differences.

Impact: For VA to realize its vision of being a world leader in providing lifelong, gender-sensitive amputation care, assessing prosthetic and functional outcomes among women is critical, as is understanding the factors that may negatively and positively contribute to women's prosthetic and functional outcomes. This study would significantly expand the evidence base for women Veterans with LEA and produce information that would inform improvements in clinical care for this population.

ELIGIBILITY:
Inclusion Criteria:

Aim 1 (prosthetic prescription, device types, and time to prescription using administrative data):

* Male or female Veteran with a first major lower extremity amputation performed in VA Medical Center between FY05 and FY18, regardless of etiology.
* Amputation will be determined based on having an inpatient or outpatient procedure code for a major lower extremity amputation (ICD-9 CM 84.13-84.19; ICD-10 codes and CPT codes also assessed but not detailed here because of space limitations).
* Patients will need to have had at least one VHA outpatient encounter in the 24 months prior to their amputation.

Aim 2 (qualitative interviews with women):

* Women Veteran VHA patients who have had a major lower extremity amputation, self-reported receiving a prescription for a prosthesis at least 12 months prior, and alive.

Aim 3 (prosthetic use, satisfaction, and functional mobility using survey data):

* Men and women Veteran VHA patients who have had a major lower extremity amputation, self-reported prescription for a prosthesis at least 12 months prior, and be alive.

Exclusion Criteria:

Aim 1 (prosthetic prescription, device types, and time to prescription using administrative data):

* prior major amputation
* unable to ambulate prior to amputation , including spinal cord injury, paraplegia, hemiplegia, or quadriplegia
* dementia
* hemipelvectomy or hip disarticulation
* ankle disarticulation
* bilateral amputation or not definitive
* death in the 3 weeks after index amputation

Aim 2 (Qualitative interviews with women):

* Specified based on eligibility criteria above.

Aim 3 (prosthetic use, satisfaction, and functional mobility using survey data):

* Specified based on eligibility criteria above.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Specified above. However, gender-based criteria ONLY applies to Aim 2 interviews. For Aim 1 administrative data and Aim 3 surveys, both men and women will be included.
Study Population: VHA patients - national sample
Sampling Method: Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Prosthetic prescription rate | 12-months post first major amputation
  Prosthetic prescription determined based on data in VA electronic medical records Sample will include those with an amputation between October 2004 (start of FY2005) and September 2018 (end of FY2018)
Use of prosthesis | July 2020-December 2021
  Orthotics and Prosthetics Users' Survey (OPUS) - 2 items Item 1: Hours per day of wear time for prosthesis Item 2: Hours per day of walking on prosthesis

SECONDARY OUTCOMES:
Functional satisfaction with prosthesis | July 2020-December 2021
  Trinity Amputation and Prosthesis Experiences Scales (TAPES) Satisfaction subscale Functional satisfaction (5 items) - score range: 5-15 (higher score = more satisfied)
Overall satisfaction with prosthesis | July 2020-December 2021
  Trinity Amputation and Prosthesis Experiences Scales (TAPES) Satisfaction subscale Overall satisfaction (1 item) - score range: 0 (not at all satisfied) to 10 (very satisfied)
Aesthetic satisfaction with prosthesis | July 2020-December 2021
  Trinity Amputation and Prosthesis Experiences Scales (TAPES) Satisfaction subscale Aesthetic satisfaction (3 items) - score range: 3-9 (higher score = more satisfied)
Functional mobility | July 2020-December 2021
  Prosthetic Limb Users Survey (PLUS-M)
Health-related quality of life | July 2020-December 2021
  PROMIS Scale V1.2 - Global Health which has two subscales - Global Physical Health (range 16.2-67.7) and Global Mental Health (21.2-67.6) Higher scores indicate better health Mean=50, Standard Deviation=10

OTHER OUTCOMES:
Amputee Single Item Mobility Measure (AMPSIMM) | July 2020-December 2021
  Scores range from 0 (less mobility) to 6 (greater mobility)

CONTACTS AND LOCATIONS:
Overall Officials: Alyson J. Littman, PhD MPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared.
Supporting Information: Study Protocol, ICF
Access Criteria: Subject to IRB approval, de-identified data will be released to a local VAPSHCS and/or national VA research data repository for release to non-VA protocols. The VA research data repository administrator will be responsible for reviewing and responding to requests to release data to non-VA requesters. A data use agreement compliant with VHA Handbooks 1200.12 and 1605.1 will be required between VHA and the requester. Review and approval by VA privacy officer is required prior to disclosure.

REFERENCES:
- [Result] Lehavot K, Young JP, Thomas RM, Williams RM, Turner AP, Norvell DC, Czerniecki JM, Korpak A, Littman AJ. Voices of Women Veterans with Lower Limb Prostheses: a Qualitative Study. J Gen Intern Med. 2022 Sep;37(Suppl 3):799-805. doi: 10.1007/s11606-022-07572-8. Epub 2022 Sep 1. PMID 36050521

DOCUMENTS (1):
  • Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT03733054/ICF_000.pdf